CLINICAL TRIAL: NCT02555137
Title: Early Non-invasive Detection of CTEPH After Pulmonary Embolism - The InShape-2 Study
Brief Title: Early Non-invasive Detection of CTEPH After Pulmonary Embolism
Acronym: InShape2
Status: Completed | Type: Observational
Sponsor: Leiden University (Other)
Responsible Party: Principal Investigator, Erik Klok, principal investigator, Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Other Study IDs: NL54450.058.15
Record Dates: First submitted 2015-09-15; First posted 2015-09-21 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
Keywords: chronic thromboembolic pulmonary hypertension; pulmonary embolism; pulmonary hypertension; screening; echocardiography
MeSH Terms: conditions — Pulmonary Embolism; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- outcome cohort study: 'prediction score' and 'rule-out criteria'
  Interventions: Other: 'prediction score' and 'rule-out criteria'

INTERVENTIONS:
Other: 'prediction score' and 'rule-out criteria' — The combination of the 'prediction score' and the 'rule-out criteria' constitutes an accurate follow-up after PE aimed at diagnosing CTEPH in early stages.

SUMMARY:
This is a prospective, international, multicenter outcome cohort study. This study starts at the moment patients visit the outpatient clinic 3 to 6 months after a diagnosis of acute PE as part of routine medical care. If patients consent to study participation, the CTEPH clinical prediction score will be calculated. CTEPH is considered to be not present in patients with a low probability (≤6 points) and no symptoms suggestive of CTEPH, i.e. dyspnea on exertion, edema, newly developed palpitations, syncope or chest pains.The remaining patients with either high probability (>6 points) or who report symptoms that may be associated with CTEPH will be subjected to the 'rule-out criteria'. CTEPH will be assumed not present in patients with an age- and gender dependent normal NT-proBNP level (as defined by the assay's manufacturer), in the absence of any of the 3 ECG criteria. Patients who have an abnormal result from the 'rule-out criteria' will be referred for transthoracic echocardiography. All echocardiograms will be performed according to a predefined standardized protocol.

In case of echocardiographic intermediate or high probability of PH, patients will be referred for further diagnostic work-up of suspected CTEPH starting with perfusion lung scan or VQ-scan and right heart catheterization, of which the results will be discussed by an independent interdisciplinary working group of PH specialists, to ensure optimal diagnostic management. This latter diagnostic work-up of an abnormal echocardiograph lies within the setting of standard medical care.

All patients who were not diagnosed with pulmonary hypertension of any origin, or with NYHA class III or IV heart failure due to left ventricular systolic dysfunction, left ventricular diastolic dysfunction or significant valvular lesions, will be followed for a total of 2 years from the index PE diagnosis. During that period, the study protocol will not interfere with standard patient care, allowing diagnostic tests as deemed indicated by the treating physician including echocardiography in case of new respiratory symptoms. At the end of the follow-up period, all patients will be subjected to a second echocardiography that will be handled according to the above stated procedures to evaluate the presence of CTEPH.

DETAILED DESCRIPTION:
This is a prospective, international, multicenter outcome cohort study. This study starts at the moment patients visit the outpatient clinic 3 to 6 months after a diagnosis of acute PE as part of routine medical care. If patients consent to study participation, the CTEPH clinical prediction score will be calculated. This score consists of 6 variables that should be assessed at the time of PE diagnosis: unprovoked PE (+6 points), known hypothyroidism (+3 points), diagnostic delay >2 weeks (+3 points), right ventricular dysfunction on computed tomography pulmonary angiography (CTPA) or echocardiography (+2 points), known diabetes mellitus (-3 points) and thrombolytic therapy or embolectomy for the acute PE event (-3 points) CTEPH is considered to be not present in patients with a low probability (≤6 points) and no symptoms suggestive of CTEPH, i.e. dyspnea on exertion, edema, newly developed palpitations, syncope or chest pains. The remaining patients with either high probability (>6 points) or who report symptoms that may be associated with CTEPH will be subjected to the 'rule-out criteria'. CTEPH will be assumed not present in patients with an age- and gender dependent normal NT-proBNP level (as defined by the assay's manufacturer), in the absence of these 3 ECG criteria: 1) rSR' or rSr' pattern in lead V1, 2) R:S >1 in lead V1 with R >0.5mV and 3) QRS axis >90o. Patients who have an abnormal result from the 'rule-out criteria' will be referred for transthoracic echocardiography. All echocardiograms will be judged by the echocardiographic criteria for suspected PH according to the 2015 ESC guidelines.

In case of echocardiographic intermediate or high probability of PH, patients will be referred for further diagnostic work-up of suspected CTEPH starting with perfusion lung scan or VQ-scan and right heart catheterization, of which the results will be discussed by an independent interdisciplinary working group of PH specialists, to ensure optimal diagnostic management. This latter diagnostic work-up of an abnormal echocardiograph lies within the setting of standard medical care.

All patients who were not diagnosed with pulmonary hypertension of any origin, or with NYHA class III or IV heart failure due to left ventricular systolic dysfunction, left ventricular diastolic dysfunction or significant valvular lesions, will be followed for a total of 2 years from the index PE diagnosis. During that period, the study protocol will not interfere with standard patient care, allowing diagnostic tests as deemed indicated by the treating physician including echocardiography in case of new respiratory symptoms. At the end of the follow-up period, all patients will be subjected to a second echocardiography that will be handled according to the above stated procedures to evaluate the presence of CTEPH.

ELIGIBILITY:
Inclusion Criteria:

* All patients with an objectivated first or recurrent diagnosis of symptomatic acute PE, who have been treated for at least three months with therapeutically dosed anticoagulant therapy according to current guidelines;
* Signed and dated informed consent of the subject available before the start of any specific study procedures;
* Age ≥18 years;

Exclusion criteria:

* Known CTEPH or PH;
* Known (i.e. echocardiographic confirmed) NYHA class III or IV chronic heart failure due to left ventricular systolic dysfunction, left ventricular diastolic dysfunction or significant valvular lesions;
* Severe renal failure (eGFR <15 ml/min) or renal replacement therapy;
* Medical or psychological condition that would not permit completion of the study or signing of informed consent, including life expectancy less than six months, or unwillingness to sign informed consent;
* Non-compliance or inability to adhere to treatment or to the follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients treated for objectivated symptomatic acute PE
Sampling Method: Non-Probability Sample
Enrollment: 424 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
The accuracy of the screening algorithm to detect CTEPH, as reflected by the 2-year incidence of confirmed CTEPH in patients in whom CTEPH was initially considered not present based on the 'risk stratification score' and the 'rule out criteria'. | 2-year follow-up
  The primairy endpoint is to evaluate the diagnostic accuracy of a CTEPH screening program based on the 'risk stratification score' and the 'rule out criteria'.

SECONDARY OUTCOMES:
The cumulative incidence and incidence rate of CTEPH in the total study population with corresponding 95% confidence interval | 2-year follow-up
  The cumulative incidence and incidence rate of CTEPH in the total study population will be calculated with corresponding 95% confidence interval
Feasibility of the screening algorithm, the number of necessary echocardiograms at baseline and the number of relevant echocardiographic findings at baseline, i.e. those that require treatment | 2-year follow-up
  number of necessary echocardiograms at baseline and the number of relevant echocardiographic findings at baseline, i.e. those that require treatment
3 Cost-effectiveness of the screening algorithm: a study-based cost-effectiveness analysis (CEA: diagnostic costs per early CTEPH diagnosis) and a model-based cost-utility analysis (CUA: societal costs per QALY). | 2-year follow-up
  cost-effectiveness of the strategy for standardized follow-up after PE aimed at diagnosing CTEPH in early stages.The economic evaluation will include a study-based cost-effectiveness analysis (CEA: diagnostic costs per early CTEPH diagnosis) and a model-based cost-utility analysis (CUA: societal costs per QALY).
incremental diagnostic accuracy of electrocardiographically derived ECG-vectoranalysis on top of the manual ECG assessment by comparing the c-statistics and reclassification numbers between the manually and automatically assessed ECG parameters | 2-year follow-up
  The additional diagnostic accuracy of the electrocardiographically derived ECG-VCG will be assessed by comparing the c-statistics and reclassification numbers between the manually and automatically assessed ECG parameters in the algorithm.
Inter-observer variability in the measurement of the RV/LV ratio on computed tomography pulmonary angiography (CTPA) expressed as the kappa-value of the ventricular dimension measurements by two independent researchers. | 2-year follow-up
  Determination of the inter-observer variability in the measurement of the RV/LV ratio on computed tomography pulmonary angiography (CTPA).

CONTACTS AND LOCATIONS:
Overall Officials: F.A. Klok, MD PhD, Principal Investigator — Department of Thrombosis and Hemostasis LUMC Leiden
Locations (5):
- UZ Leuven, Leuven, Belgium
- Netherlands (3):
  - VUmc, Amsterdam
  - LUMC, Leiden
  - Haga, The Hague
- medical university of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Klok FA, Tesche C, Rappold L, Dellas C, Hasenfuss G, Huisman MV, Konstantinides S, Lankeit M. External validation of a simple non-invasive algorithm to rule out chronic thromboembolic pulmonary hypertension after acute pulmonary embolism. Thromb Res. 2015 May;135(5):796-801. doi: 10.1016/j.thromres.2014.12.009. Epub 2014 Dec 13. PMID 25746363
- [Result] Klok FA, Surie S, Kempf T, Eikenboom J, van Straalen JP, van Kralingen KW, van Dijk AP, Vliegen HW, Bresser P, Wollert KC, Huisman MV. A simple non-invasive diagnostic algorithm for ruling out chronic thromboembolic pulmonary hypertension in patients after acute pulmonary embolism. Thromb Res. 2011 Jul;128(1):21-6. doi: 10.1016/j.thromres.2011.03.004. Epub 2011 Mar 30. PMID 21450333
- [Derived] Fabyan KD, Holley AB. Postpulmonary embolism syndrome. Curr Opin Pulm Med. 2021 Sep 1;27(5):335-341. doi: 10.1097/MCP.0000000000000789. PMID 34127618